CLINICAL TRIAL: NCT06124937
Title: Evaluating the Role of EMpagliflozin on the Rate of Post-Operative Atrial Fibrillation in Patients Undergoing Coronary Artery Bypass Graft Surgery: a Double-blind Placebo-controlled Randomized Clinical Trial
Brief Title: Empagliflozin to Prevent Post-Operative Atrial Fibrillation
Acronym: EMPOAF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rajaie Cardiovascular Medical and Research Center (Other)
Collaborators: Tehran Heart Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRCT20230110057098N1
Record Dates: First submitted 2023-10-23; First posted 2023-11-09 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Post-operative Atrial Fibrillation; CABG
Keywords: Atrial Fibrillation; CABG; Cardiac surgery; Empagliflozin; Post-operative AF; SGLT2 inhibitors
MeSH Terms: conditions — Atrial Fibrillation | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Two arms, parallel-group, phase 3, randomized, double-blind, placebo-controlled trial with allocation sequence concealment and blinded endpoint adjudication on 492 patients
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither the participants nor the researchers know which treatment or intervention patients are receiving
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive a 10 mg tablet of empagliflozin once a day from 3 days before surgery until discharge from the hospital.
  Interventions: Drug: Empagliflozin 10 MG
- Comperator (Placebo Comparator): The comparator group will receive a matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 MG — The intervention group will receive a 10 mg tablet of empagliflozin once a day from 3 days before surgery until discharge from the hospital.
  Arms: Intervention group
Drug: Placebo — The comparator group will receive a matching placebo from 3 days before surgery until discharge from the hospital.
  Arms: Comperator

SUMMARY:
This is an interventional, double-blind, placebo controlled, multicenter, randomized clinical trial with allocation sequence concealment and blinded endpoint adjudication. The goal of present study is to investigate if periprocedural administration of 10 mg once daily empagliflozin, a sodium-glucose cotransporter-2 inhibitor (SGLT2I), can reduce the incidence of post-operative atrial fibrillation and/or atrial flutter in patients with chronic coronary syndrome scheduled for isolated CABG. This trial will be conducted in two referral teaching cardiology hospitals in Tehran. 492 adult patients who are scheduled for elective isolated coronary artery bypass graft (CABG) surgery will be randomly assigned to one of the groups of intervention (empagliflozin 10 mg daily) or placebo starting 3 days before surgery until discharge.

DETAILED DESCRIPTION:
Study aim: Evaluating the role of empagliflozin on the rate of postoperative atrial fibrillation in comparison with placebo Design: Two arms, parallel-group, phase 3, randomized, double-blind, placebo-controlled trial on 492 patients Settings and conduct: Recruitment site: Tehran Heart Center and Rajaie Cardiovascular Medical and Research Center For blinding, the drug or placebo will be given to the ward based on the patient's code in the randomization system For monitoring, the blood samples for creatinine, sodium, potassium, and fasting blood sugar along with clinical evaluations will be given on day 0 and daily thereafter (max= 30 days) in specific wards and will be compared at the end of any atrial fibrillation lasting longer than 30 seconds based on 24-hour 12-lead ECG monitoring will be accepted as atrial fibrillation After entering the study, the patients are placed in one of two groups, sample and control; in the sample group, they are treated with the usual treatment regimen plus empagliflozin at a dose of 10 mg during the hospitalization period. Patients in the control arm will receive a matching placebo.

ELIGIBILITY:
Inclusion criteria

* Adult patients (≥18 years) who are candidates for isolated CABG
* Patients who provided written informed consent and are willing to participate in the study

Exclusion criteria

* History of type Ⅰ or Ⅱ diabetes mellitus
* History of ketoacidosis
* History of atrial fibrillation or flutter
* History of recurrent UTI
* SGLT2I or any other oral hypoglycemic medications used due to other indications
* Patients with acute kidney injury (45)
* Severe hepatic disease (Child-Pugh score C)
* Patients with Estimated Glomerular Filtration Rate (eGFR) < 30 mL/min/1.73m2
* Patients who are candidates for emergent CABG
* Patients with unstable hemodynamic state
* Patients with positive urine culture, urinary symptoms (frequency, dysuria, hesitancy), and asymptomatic bacteriuria
* Patients who are enrolled in other clinical trials
* Patients with a history of drug-sensitive reactions to SGLT2I
* Pregnancy or lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of POAF | From CABG until discharge from the intensive care unit (at least 72 hours and maximum 30 days)
  Incidence of new-onset postoperative atrial fibrillation (AF) and/or atrial flutter (AFL), defined as any adjudicated documented AF or AFL of at least 30 seconds duration and documented by Holter ECG monitoring during the admission time in the ICU (at least 72 hours and maximum 30 days).

SECONDARY OUTCOMES:
Composite Incidence of all arrhythmias leading to hemodynamic instability | From CABG until discharge from the hospital (maximum 30 days).
  Defined as any adjudicated documented tachy- or bradyarrhythmia of at least 30 seconds duration and documented by rhythm strips or 12-lead ECG leading to hemodynamic instability during the admission time. Ventricular tachycardia (VT) of at least 30 seconds duration and documented by rhythm strip or 12-lead ECG.
  Ventricular fibrillation (VF) of at least 30 seconds duration and documented by rhythm strip or 12-lead ECG
Incidence of post-operative acute kidney injury | From CABG until 7th post-operation day.
  Defined as the presence of either the increase in serum creatinine by ≥ 0.3 mg/dl (≥ 26.5 µmol/l) within 48 hours; or an increase in serum creatinine to ≥ 1.5 times baseline, which is known or presumed to have occurred within the prior 7 days; or urine volume < 0.5 ml/kg/h for 6 hours based on the KDIGO definition of AKI
Need for vasopressor/inotrope | From CABG until discharge from the intensive care unit (maximum 30 days).
  Defined as cumulative vasopressor index and the amount of average daily inotrope dose during the admission time in the ICU
Duration of hospitalization | From CABG until discharge from the hospital.
  Defined as number of days a patient stay at the hospital
All-cause mortality | From CABG until 30th post-operation day.
  Defined as adjudicated 30-day mortality, including cause-specific mortality: cardiac arrhythmic, cardiac non-arrhythmic, and non-cardiovascular.
Incidence of life-threatening infections | From CABG until discharge (maximum 30 days).
  Defined as any adjudicated laboratory and clinically confirmed systemic infection that necessitate the administration of parenteral broad spectrum antibiotics
Incidence of genitourinary tract infections | From CABG until discharge from the hospital (maximum 30 days).
  Defined as any adjudicated laboratory and clinically confirmed genitourinary tract infection including cystitis, pyelonephritis, prostatitis, urethritis, and vaginitis
Incidence of hypoglycemia | From CABG until discharge from the hospital (maximum 30 days).
  Defined as serum blood sugar ≤ 70 mg/dL (≤ 3.9 mmol/L)
Incidence of ketoacidosis | From CABG until discharge from the hospital (maximum 30 days).
  Defined as blood pH ≤ 7.3, serum bicarbonate less than 15 mEq/l, and presence of ketonemia or ketonuria
Incidence of clinically-diagnosed ischemic stroke | From CABG until 30th post-operation day.
  Defined as the sudden loss of blood circulation to an area of the brain that has been confirmed with appropriate diagnostic imaging (Brain CT/MRI)
Composite incidence of arterial and venous thrombosis | From CABG until 30th post-operation day.
  Defined as adjudicated arterial thrombosis (including Type I MI and peripheral arterial thrombosis) and venous thrombosis (including DVT and PE) confirmed with appropriate diagnostic tools
Need for renal replacement therapy | From CABG until discharge from the intensive care unit (maximum 30 days).
  defined as treatment with any forms of dialysis (hemodialysis, hemodiafiltration, and peritoneal dialysis), hemofiltration, and renal transplantation

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - Tehran Heart Center, Tehran
  - Rajaie Cardiovascular Medical & Research Center, Tehran

IPD SHARING:
Plan to Share IPD: Undecided